CLINICAL TRIAL: NCT03312049
Title: Relationship Between Maternal Exposure to Mycotoxins, Birth Outcomes and Stunting in Infants: A Birth Cohort Study in Nepal
Brief Title: Aflatoxin Birth Cohort Study Nepal (AflaCohort)
Acronym: AflaCohort
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Collaborators: Helen Keller International (Other); Patan Academy of Health Sciences (Other); Purdue University (Other); Government of Nepal (Unknown); Nepalgunj Medical College (Unknown)
Responsible Party: Principal Investigator, Patrick Webb, Alexander McFarlane Professor of Nutrition, Tufts University
Other Study IDs: USAID AID-OAA-G-14-0000
Record Dates: First submitted 2017-09-11; First posted 2017-10-17 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Stunting; Birth Weight; Birth Length; Height for Age; Linear Growth Failure
Keywords: Aflatoxin B1; Aflatoxin M1; Aflatoxin; Mycotoxin; Stunting; Linear growth; Pregnancy; Birth outcomes; Nepal
MeSH Terms: conditions — Growth Disorders; Birth Weight; Failure to Thrive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum aflatoxin B1-lysine adduct levels Breast milk aflatoxin M1 levels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study focuses on the causal relationship between mycotoxin exposure (particularly aflatoxin B1), birth outcomes, and height for age among young children in Nepal. Previous studies have shown a strong association of stunting with mycotoxin exposure yet causality has not been proven. Thus, this study will provide a better understanding of the association between maternal and/or early life mycotoxin exposure (rates in the blood and breast milk) and infant and young child growth. This information is essential if we are to more fully understand and effectively address the high rates of stunting in Asia.

DETAILED DESCRIPTION:
In 2012, a research prioritization meeting organized by IFPRI and the Bill and Melinda Gates Foundation on food-borne toxins concluded, "While there is solid association of stunting with exposure to mycotoxins, the causality has not been proven and the percentage of stunting attributable to mycotoxins in general or to specific mycotoxins is not known." (IFPRI/BMGF 2012) In other words, the extent of the problem, although widely suspected, has been poorly documented and the biological mechanisms thought to be involved remain poorly understood.

To contribute to a better understanding of the mycotoxin-stunting relationship, the Feed the Future Feed the Future Nutrition Innovation Lab-Asia proposes to explore the impact of mycotoxins, with a focus on mycotoxins on child nutrition in Nepal. Through its PoSHAN study, the Nutrition Innovation Lab-Asia is currently undertaking research in Nepal in collaboration with the Child Health Division of the Ministry of Health and Population and multiple local partners on how investments in agriculture can achieve significant impacts on maternal and child nutrition, and on demonstrating how large-scale programs best incorporate such evidence into cost-effective multi-sectoral interventions. Adding a study component on food safety (mycotoxin contamination of the food supply) will significantly enhance our understanding of nutrition outcomes linked to investments in agriculture. As noted by participants of the IFPRI/BMGF (2012) meeting, "only 35% of stunting of children can be attributed to known factors". This leaves room for research to uncover other suspected contributors to the world's huge nutrition problems, which could then lead testable recommendations for innovative interventions to address newly identified factors. The team will assess current mycotoxin risk so that potential mitigation strategies can be developed.

Given the significant statistical associations shown between mycotoxin exposure in children and height gain in infants and young children, the Nutrition Innovation Lab-Asia will undertake an mycotoxin birth cohort study to further the understanding of the causal relationship between past and current mycotoxin exposure (maternal and infant), birth outcomes and length-for-age in Nepali infants and young children. The study will also seek to validate the use of low cost data collection methods (e.g. dried blood spots versus venous blood samples) for mycotoxin analysis.

The specific aims of this study are:

1. To examine the relationship of maternal mycotoxin exposure in pregnancy and birth outcomes, including infant birth weight.
2. To examine the relationship of exposure to mycotoxin of infants through breast milk and their linear growth.
3. To examine the relationship of exposure to mycotoxin through complementary feeding and linear growth.
4. To enumerate the relative contributions of maternal and infant mycotoxin exposures in impairing linear growth, controlling for other potential explanatory factors.

Controlling for factors such as diet, maternal education, maternal height and BMI, household socio-economic status, infections and inflammation, and other elements such as storage patterns, knowledge of food contaminants and mitigation practices, the specific hypotheses of this study are:

1. There is an incremental effect of in utero, lactation and complementary feeding mycotoxin exposures on rate of length gain and stunting outcomes for age Z-scores in children at 2 year of age.
2. Maternal exposure to mycotoxins will be significant predictor of birth weight in infants, thereby being a significant contributor to the burden of stunting at 2 years of age.
3. Exposure to mycotoxins through breast milk before 6 months of age along with continued exposure through both breast milk and complementary foods (after 6 months of age) is a significant contributor to the burden of stunting at 2 years of age.
4. Improper farm management, food processing and storage practices are significantly related to higher levels of serum mycotoxins in the blood of mothers and their children.
5. Knowledge of the problem of food-borne contaminants is associated with improved food processing and storage practices.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and adolescent girls (less than 30 weeks gestation)
* Aged 16-49 years
* Living in the study area
* Intends to reside in the study area through the study period
* Intends to deliver in the study area
* Provides informed consent herself or through a legal guardian
* Live Birth
* Single Birth

Exclusion Criteria:

* Severely malnourished mother <17.5 cm
* Severely anemic mother hemoglobin<7 g/dL
* Pregnancy induced hypertension
* Congenital anomalies
* Very low birth weight <1500 g
* Sepsis
* Respiratory distress syndrome
* Severe malnutrition infant ≤-3 WFH z-score (3 months), <11.5 cm MUAC or edema
* Severe anemia infant (hemoglobin<7 g/dL)
* Fetal loss
* Early termination of pregnancy
* Still births
* Infant death
* Relocation of household

Ages: 16 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Pregnant women and adolescent girls
Study Population: All pregnant women and adolescent girls aged 16-49 years and living in the study areas will be invited to join the study. Women who are less than 30 weeks into their gestation will be eligible to participate if their expected delivery date falls within the enrollment period.
Sampling Method: Non-Probability Sample
Enrollment: 1675 (Actual)
Dates: Start 2015-07-06 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Height for Age Z-scores (HAZ) | Measured at birth and when infant turns 3, 6, 9, 12, 18 and 24 months of age
  Height for Age Z-scores based on the World Health Organization's 2006 Child Growth Standards, HAZ < -6 and > 6

SECONDARY OUTCOMES:
Aflatoxin M1 (breast milk) | Measured when infant is 3 months of age
  High-performance liquid chromatography (HPLC) method used to measure ng aflatoxin M1 per liter of breast milk (ng/L)
Low birth weight | Measured at birth
  < 2500 g
Aflatoxin B1 (serum) | Measured during pregnancy
  High-performance liquid chromatography (HPLC) method used to measure pg aflatoxin B1-lysine adducts per mg albumin
Change in infant aflatoxin B1 | Measured when infant turns 3, 6, 12 and 18 months of age
  High-performance liquid chromatography (HPLC) method used to measure pg aflatoxin B1-lysine adducts per mg albumin
Fumonisin B, Deoxynivalenol (DON) (urine) | Measured when infant turns 18 months of age
  High-performance liquid chromatography (HPLC)
Ochratoxin A (serum) | Measured when infant turns 18 months of age
  High-performance liquid chromatography (HPLC)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Webb, PhD, Principal Investigator — Tufts University; Kedar P Baral, MD, Principal Investigator — Patan Academy of Health Sciences; Shibani Ghosh, PhD, Principal Investigator — Tufts University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lamichhane A, Webb P, Andrews-Trevino J, Pokharel A, Acharya S, Shrestha R, Davis D, Baral K, Wang JS, Xue K, Paudel K, Ghosh S. Dietary determinants of aflatoxin B1-lysine adduct among infants in Nepal. Eur J Clin Nutr. 2022 Nov;76(11):1557-1565. doi: 10.1038/s41430-022-01142-1. Epub 2022 Apr 20. PMID 35444268
- [Derived] Andrews-Trevino JY, Webb P, Shively G, Kablan A, Baral K, Davis D, Paudel K, Shrestha R, Pokharel A, Acharya S, Wang JS, Xue KS, Ghosh S. Aflatoxin exposure and child nutrition: measuring anthropometric and long-bone growth over time in Nepal. Am J Clin Nutr. 2021 Apr 6;113(4):874-883. doi: 10.1093/ajcn/nqaa397. PMID 33677532
- [Derived] Andrews-Trevino JY, Webb P, Shively G, Rogers BL, Baral K, Davis D, Paudel K, Pokharel A, Shrestha R, Wang JS, Ghosh S. Relatively Low Maternal Aflatoxin Exposure Is Associated with Small-for-Gestational-Age but Not with Other Birth Outcomes in a Prospective Birth Cohort Study of Nepalese Infants. J Nutr. 2019 Oct 1;149(10):1818-1825. doi: 10.1093/jn/nxz122. PMID 31198947